CLINICAL TRIAL: NCT00762268
Title: Intermittent-Dose Oral SAMe (S-adenosyl-L-methionine) in Persistent and Treatment-Refractory Bipolar Depression: A Double-Blind Pilot Trial With an Optional Open-label Follow-up
Brief Title: A Trial of SAMe for Treatment-Resistant Bipolar Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Beth L. Murphy MD, PhD, Principal Investigator, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-P-000276
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Bipolar Disorder; Depression; Bipolar Depression
Keywords: SAMe; alternative treatments; bipolar disorder; depression; bipolar depression; treatment-resistant depression
MeSH Terms: conditions — Bipolar Disorder; Depression; Depressive Disorder, Treatment-Resistant | interventions — S-Adenosylmethionine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SAMe (Experimental): SAMe: SAMe tablets will be administered intermittently and in steadily increasing dosages. Subjects will receive oral SAMe for only 3 days per week, followed by a 4 day "rest-period", before the next dosage increase. SAMe dosage will be progressively increased each week to a maximum of 1600 mg per day over a 4-week period.
  Interventions: Drug: SAMe
- placebo (Placebo Comparator): Placebo: Placebo SAMe tablets will be administered intermittently and in steadily increasing dosages. Subjects will receive oral pills for only 3 days per week, followed by a 4 day "rest-period", before the round. The apparent dosage will be progressively increased each week to mimic a maximum of 1600 mg per day over a 4-week period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAMe — SAMe tablets will be administered intermittently and in steadily increasing dosages. Subjects will receive oral SAMe for only 3 days per week, followed by a 4 day "rest-period", before the next dosage increase. SAMe dosage will be progressively increased each week to a maximum of 1600 mg per day over a 4-week period.
  Other Names: S-adenosyl-L-methionine
  Arms: SAMe
Drug: Placebo
  Arms: placebo

SUMMARY:
S-adenosyl-L-methionine (SAMe) is a dietary supplement with antidepressant properties. SAMe's mechanism of action remains unclear, but it appears to be distinct from that of conventional antidepressants. The purpose of this study is to examine the effect of these properties on the mood of bipolar subjects with persistent major depression that has been unresponsive to standard pharmacotherapy.

DETAILED DESCRIPTION:
Depression in bipolar disorder is a significant source of disease-related debility; with bipolar individuals typically spending three fold as much time depressed as manic or hypomanic. Clinicians treating bipolar disorder often struggle to provide relief from depressive symptoms that are more often treatment resistant than in unipolar depression. To complicate matters further, the risk/benefit ratio of currently available antidepressants is a source of debate within the field of psychiatry.

S-adenosyl-L-methionine (SAMe) is a dietary supplement with well-established antidepressant properties. SAMe's mechanism of action remains unclear, but it appears to be distinct from that of conventional antidepressants. The purpose of this study is to examine the effect of these properties on the mood of bipolar subjects with persistent major depression that has been unresponsive to standard pharmacotherapy.

An unusual aspect of the current study design is the schedule of SAMe dosing. SAMe tablets will be administered intermittently and in steadily increasing dosages. The purpose of this gradual and intermittent dosage titration is to lessen the risk of antidepressant-induced mania by seeking the minimum effective oral dose of SAMe.

ELIGIBILITY:
Inclusion Criteria:

* bipolar disorder
* depressed for 3-12 months
* mood unresponsive to at least 2 treatments
* currently on mood stabilizer at therapeutic doses

Exclusion Criteria:

* history of mania while on adequate mood stabilizer
* rapid cycling bipolar disorder
* previous use of SAMe during current episode
* unstable medical illness including parkinson's disease
* methotrexate use
* pregnancy
* substance abuse/dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth L Murphy, MD, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Result] Murphy BL, Babb SM, Ravichandran C, Cohen BM. Oral SAMe in persistent treatment-refractory bipolar depression: a double-blind, randomized clinical trial. J Clin Psychopharmacol. 2014 Jun;34(3):413-6. doi: 10.1097/JCP.0000000000000064. No abstract available. PMID 24699040
- See also: link to hospital web site with clinical trials information — http://www.mclean.harvard.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SAMe | Placebo
Started | 12 | 11
Completed | 9 | 8
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Population: Individuals entering the treatment phase of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | SAMe | Placebo | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Scale (MADRS)
Description: Assessment of current depression symptoms using Montgomery-Asberg Depression Scale (MADRS). All 10 questions on the scale have a 0 (absent)-6(most severe) range for describing symptoms, with the total ranging from 0-60. A higher total score indicates a greater number of symptoms and higher symptom intensity, while a smaller score indicates a lesser number of symptoms and lower intensity.
Time Frame: At each weekly visit for 4 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | SAMe | Placebo
Number analyzed (Participants) | 9 | 8
units on a scale
  Baseline | 29.4 [17 to 39] | 28.3 [18 to 37]
  Week 1 | 24.7 [10 to 37] | 24.2 [11 to 37]
  Week 2 | 26.3 [16 to 46] | 23.0 [8 to 37]
  Week 3 | 23.7 [8 to 35] | 18.5 [8 to 34]
  Week 4 | 20.1 [8 to 31] | 18.1 [8 to 41]
Statistical Analysis 1: Comparison: SAMe vs Placebo; Test type: Superiority or Other; p = 1.0, Regression, Linear

2. Secondary Outcome: Hamilton Rating Scale for Depression
Description: Rating scale of depression symptoms (range 0-50). A higher total score indicates a greater number of symptoms and higher symptom intensity, while a smaller score indicates a lesser number of symptoms and lower intensity.
Time Frame: 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SAMe | Placebo
Number analyzed (Participants) | 7 | 6
units on a scale | 11.9 (7.6) | 7.3 (0.9)
Statistical Analysis 1: Comparison: SAMe vs Placebo; Change from intake scores; Test type: Other; p = 0.05, Chi-squared

3. Secondary Outcome: Young Mania Rating Scale
Description: Rating scale for manic symptoms (range 0-60). A higher total score indicates a greater number of symptoms and higher symptom intensity, while a smaller score indicates a lesser number of symptoms and lower intensity.
Time Frame: 6-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SAMe | Placebo
Number analyzed (Participants) | 7 | 6
units on a scale | 2.8 (2.0) | 1.8 (0.5)
Statistical Analysis 1: Comparison: SAMe vs Placebo; Test type: Other; p = 0.05, Chi-squared

ADVERSE EVENTS:
Arm/Group | SAMe | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 1/9 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAMe (N=9) | Placebo (N=8)
Auditory Hallucinations (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No